CLINICAL TRIAL: NCT07300345
Title: Liver Affection in Pregnant Women at Sohag University Hospitals
Brief Title: Liver Affection in Pregnant Women at Sohag University Hospital
Acronym: LAIPWASUH
Status: Not yet recruiting | Type: Observational
Sponsor: Eman Ashraf Saad Ahmed (Other)
Responsible Party: Sponsor-Investigator, Eman Ashraf Saad Ahmed, resident doctor, tropical medicine and gastroentrology, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med--25-11-4MS
Record Dates: First submitted 2025-11-28; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Liver Biomarkers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- all pregnant women attending sohag university hospitals for liver disease assessment: Participants in this group will undergo a single assessment during their hospital visit. This includes history taking, brief medical history, and collecting routine laboratory and imaging results. No additional procedures or intervention will be performed specifically for this study. The purpose is estimate prevalence of liver diseases in pregnant women

SUMMARY:
This study investigates the prevalence, causes, and clinical outcomes of liver disorders among pregnant women attending Sohag University Hospital. It aims to identify the most common hepatic conditions occurring during pregnancy, evaluate their impact on maternal and fetal health, and assess the effectiveness of current diagnostic and management approaches. By analyzing clinical data, laboratory findings, and pregnancy outcomes, the study highlights the importance of early detection and proper management of liver diseases to reduce associated complications and improve overall maternal-fetal prognosis.

DETAILED DESCRIPTION:
This study provides evaluation of liver disorders among pregnant women attending Sohag University Hospital. The research aims to determine the prevalence of hepatic conditions during pregnancy, classify the most common liver diseases encountered, and analyze their etiologies, clinical presentations, and laboratory characteristics. Special emphasis is placed on conditions unique to pregnancy-such as intrahepatic cholestasis of pregnancy, HELLP syndrome, and acute fatty liver of pregnancy-as well as pre-existing or coincidental liver diseases, including viral hepatitis and autoimmune hepatic disorders.

The study further examines the impact of these hepatic conditions on both maternal and fetal outcomes. . By reviewing diagnostic tools, biochemical markers, and imaging findings, the research evaluates the effectiveness of current diagnostic pathways used in the hospital setting.

ELIGIBILITY:
Inclusion Criteria:

All pregnant women >18 years old with elevated Liver enzyme levels All pregnant women >18 years old with elevated bilirubin level

Exclusion Criteria:

Pregnant women who refuse to participate in the study, Pregnant women with biliary diseases (e.g., cholangitis, cholecystitis)

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: The study population includes pregnant women attending Sohag University Hospital during the study period. Participants are women of reproductive age with a confirmed pregnancy who are diagnosed with the targeted liver disorder. Inclusion is irrespective of gestational age at diagnosis, while women with pre-existing chronic liver failure or other severe systemic illnesses are excluded. The study focuses exclusively on female participants
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in liver disease severity index | from baseline up to delivery
  Change from baseline in a standardized liver disease severity index combining biochemical and clinical measures in pregnant women. The index is computed using: serum ALT (IU/L), AST (IU/L), total bilirubin (mg/dL), albumin (g/dL), INR, and a short clinical symptom score (pruritus, jaundice, abdominal pain). Outcomes reported as absolute change and percent change in the composite score to evaluate progression or improvement of the liver disorder.